CLINICAL TRIAL: NCT04934696
Title: A Phase 1 Study to Characterize the Effects of BMS-986166 on the Pharmacokinetics of an Oral Contraceptive Containing Ethinyl Estradiol and Norethindrone in Healthy Female Participants
Brief Title: A Study to Characterize the Drug Levels of an Oral Contraceptive With and Without BMS-986166 in Healthy Female Participants of Childbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IM018-006
Record Dates: First submitted 2021-06-17; First posted 2021-06-22 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; BMS-986166
MeSH Terms: interventions — BMS-986166; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986166 + Oral contraceptive (Experimental)
  Interventions: Drug: BMS-986166; Drug: Oral contraceptive

INTERVENTIONS:
Drug: BMS-986166 — Specified dose on specified days
Drug: Oral contraceptive — Specified dose on specified days

SUMMARY:
The purpose of this study is to investigate the potential for a drug-drug interaction (DDI) when BMS-986166 and hormonal oral contraceptives are co-administered.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit: www.BMSStudyConnect.com

Inclusion Criteria:

* Nonpregnant, nonlactating Women of Childbearing Potential (WOCBP) who are healthy as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations will be eligible to participate in the study.
* Body mass index (BMI) of 18.0 to 32.0 kg/m². BMI = weight (kg)/(height[m])² for participants.
* Participant must be 18 to 45 years of age, inclusive, at the time of signing the informed consent.

Exclusion Criteria:

* Any significant acute or chronic medical illness judged to be clinically significant by the investigator and/or Sponsor Medical Monitor.
* History of any type of heart disease, including ischemia, infarction, clinically significant arrhythmias, sinus syndrome, hypertension, symptomatic orthostatic hypotension, atrioventricular block of any degree, bradycardia, syncope, clinically significant ECG abnormalities, or any congenital heart disease.
* Any acute or chronic bacterial, fungal (except history of tinea pedis or ongoing onychomycosis will not be exclusionary) or viral infection within the last 3 months prior to screening, as well as any febrile illness or viral infection within the last 3 months prior to screening, as well as any febrile illness of unknown origin within 14 days of screening.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Geometric means ratio of Cmax of NET | Up to Day 26
  Geometric means ratio of maximum observed plasma concentration (Cmax) of norethindrone (NET) when administered with versus without BMS-986166
Geometric means ratio of Cmax of EE | Up to Day 26
  Geometric means ratio of maximum observed plasma concentration (Cmax) of ethinyl estradiol (EE) when administered with versus without BMS-986166
Geometric means ratio of AUC(0-T) of NET | Up to Day 26
  Geometric means ratio of area under the plasma concentration-time curve from time zero to time of last quantifiable concentration for NET when administered with versus without BMS-986166
Geometric means ratio of AUC(0-T) of EE | Up to Day 26
  Geometric means ratio of area under the plasma concentration-time curve from time zero to time of last quantifiable concentration for EE when administered with versus without BMS-986166
Geometric means ratio of AUC(INF) of NET | Up to Day 26
  Geometric means ratio of area under the plasma concentration-time curve from time zero extrapolated to infinite time for NET administered with versus without BMS-986166
Geometric means ratio of AUC(INF) of EE | Up to Day 26
  Geometric means ratio of area under the plasma concentration-time curve from time zero extrapolated to infinite time for EE when administered with versus without BMS-986166

SECONDARY OUTCOMES:
Cmax of BMS-986166 | Up to Day 26
Cmax of BMT-121795 | Up to Day 26
Time of maximum observed plasma concentration (Tmax) of BMS-986166 | Up to Day 26
Tmax of BMT-121795 | Up to Day 26
Area under the plasma concentration-time curve in one dosing interval (AUC(TAU)) of BMS-986166 | Up to Day 26
AUC(TAU) of BMT-121795 | Up to Day 26
Tmax of EE | Up to Day 26
Tmax of NET | Up to Day 26
Terminal plasma elimination phase half-life (T-HALF) of EE | Up to Day 26
T-HALF of NET | Up to Day 26
Apparent total clearance of drug from plasma after oral administration (CLT/F) of EE | Up to Day 26
CLT/F of NET | Up to Day 26
Apparent volume of distribution at terminal phase (Vz/F) of EE | Up to Day 26
Vz/F of NET | Up to Day 26
Number of participants with Adverse Events (AEs) | Up to Day 37
Number of participants with Serious Adverse Events (SAEs) | Up to Day 37
Number of participants with clinically significant changes in laboratory values: Hematology tests | Up to Day 30
Number of participants with clinically significant changes in laboratory values: Chemistry tests | Up to Day 30
Number of participants with clinically significant changes in laboratory values: Urinalysis | Up to Day 30
Number of participants with clinically significant changes in vital signs: Body temperature | Up to Day 27
Number of participants with clinically significant changes in vital signs: Respiratory rate | Up to Day 27
Number of participants with clinically significant changes in vital signs: Blood pressure | Up to Day 27
Number of participants with clinically significant changes in vital signs: Heart rate | Up to Day 27
Number of participants with clinically significant changes in ECG parameters: PR interval | Up to Day 27
  PR interval is the time from the onset of the P wave to the start of the QRS complex
Number of participants with clinically significant changes in ECG parameters: QRS | Up to Day 27
  QRS can be defined as the electrical impulse as it spreads through the ventricles, indicating ventricular depolarization
Number of participants with clinically significant changes in ECG parameters: QT interval | Up to Day 27
  The QT interval is the time from the start of the Q wave to the end of the T wave
Number of participants with clinically significant changes in ECG parameters: QTcF | Up to Day 27
  QTcF = Corrected QT interval using the Fridericia formula. QT interval is the time from the start of the Q wave to the end of the T wave
Number of participants with physical examination abnormalities | Up to Day 27

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- West Coast Clinical Trials Global, Cypress, California, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm